CLINICAL TRIAL: NCT02031614
Title: The Immunomodulatory Effects of Phlebotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Phlebotomy-2014
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Anemia
Keywords: anemia; blood withdrawal; phlebotomy; innate immunity; Immune reponse
MeSH Terms: conditions — Anemia | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phlebotomy (Experimental): Subjects in this arm will undergo phlebotomy of 500 mL of blood.
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Phlebotomy — Withdrawal of 500 mL of whole blood.

SUMMARY:
Although phlebotomy is routinely performed in blood donors, and seemingly does not have significant health risks, it is highly relevant to know what the effect of phlebotomy is on immunity. Alterations in immunity due to phlebotomy could have beneficial effects, like the suppression of the low grade inflammatory process that contributes to atherosclerosis, but in theory could also contribute to a suppressed innate immune response that could increase the risk of infection. This is not only relevant for blood donors, but also for patients suffering from blood loss and for daily clinical practice in which blood is routinely drawn of patients for laboratory determinations.

DETAILED DESCRIPTION:
The loss of blood by haemorrhage or routine phlebotomy as performed during blood donation by healthy volunteers, has large effects on systemic iron homeostasis. The relative shortage of erythrocytes after blood loss is compensated for by increasing the production of new red cells by the bone marrow. As iron is needed for effective haemoglobin synthesis, the transport of iron to the bone marrow needs to be increased. This is accomplished by the suppression of hepcidin production in the liver. Hepcidin is the central regulator of iron homeostasis. It can regulate serum iron levels effectively by downregulating iron channel ferroportin on iron exporting cells. Hepcidin production is increased in response to inflammation en high systemic iron content, and is suppressed by increased erythrocyte production, hypoxia, anemia, and low systemic iron content. Therefore, blood loss leads to hepcidin suppression, increased release of iron into the circulation and decrease of iron stores.

Alterations in iron metabolism can have immunomodulatory effects. The intra cellular iron content in macropahges and monocytes, has shown pro-inflammatory effects in several investigations. Hepcidin is reported to have pro-inflammatory effects in some reports, and anti-inflammatory effects in others.

Although phlebotomy is routinely performed in blood donors, and seemingly does not have significant health risks, it is highly relevant to know what the effect of phlebotomy is on immunity. Alterations in immunity due to phlebotomy could have beneficial effects, like the suppression of the low grade inflammatory process that contributes to atherosclerosis, but in theory could also contribute to a suppressed innate immune response that could increase the risk of infection. This is not only relevant for blood donors, but also for patients suffering from blood loss and for daily clinical practice in which blood is routinely drawn of patients for laboratory determinations.

Objective: To assess the ex vivo cytokine production of whole blood during 28 days after phlebotomy (routine withdrawal of 500 ml of blood).

Study design: Intervention study in 10 healthy male volunteers.

Study population: 10 healthy male volunteers in the age of 18-35 years.

Intervention (if applicable): Withdrawal of 500 mL of blood at the blood bank (Sanquin, Nijmegen, The Netherlands).

Main study parameters/endpoints:

* Ex vivo cytokine production of whole blood, drawn on day -1, 0, 1, 3, 5, 7, 14, 21, 28.
* Hemoglobin, hematocrit, white blood cell count and differential
* Hepcidin
* Iron parameters (serum iron, transferrin saturation, ferritin)

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

10 healthy young male volunteers will be included in this study. The study consists of 10 visits: 1 screening visit and 9 follow-up visits. The screening visit consists of a medical history questionnaire. On day 0, Phlebotomy of 500 ml of blood will be performed at the Sanquin blood bank, Nijmegen according to normal procedures. Risks associated with phlebotomy are, discomfort during puncture, light-headedness, orthostatic hypotension, vasovagale response, and hematoma at the puncture site.

On day -1, 0, 1, 3, 5, 7, 14, 21 and 28, a volume of 7 mL of blood will be drawn by venapuncture. Associated risks are discomfort during puncture , vasovagale response, and hematoma at the puncture site.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age >18 and <36 years
* Healthy as concluded from medical history

Exclusion Criteria:

* Having donated blood to the blood bank within one year preceding phlebotomy
* Significant blood loss from trauma within one year preceding phlebotomy
* Having lost > 100 ml of blood due to any cause, within 3 months preceding phlebotomy (not counting blood withdrawn during screening visit)
* Having lost > 50 ml of blood due to any cause, within 1 month preceding phlebotomy (not counting blood withdrawn during screening visit)
* Having lost >20 ml blood due to any cause, within 1 week preceding phlebotomy (not counting blood withdrawn during screening visit)
* Family history of thallasemia, sickle cell disease, hereditary hemochromatosis, or iron refractory iron deficiency anemia
* Signs of history of infection within 2 weeks preceding phlebotomy
* History of frequent vasovagal response

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
ex vivo TNF-afpha production of whole blood in reponse to incubation with E. Coli LPS | 1 day before till 28 days after phlebotomy
  Blood will be drawn on day -1, 0, 1, 3, 5, 7, 14, 21 and 28 after phlebotomy, to assess ex vivo cytokine production.

SECONDARY OUTCOMES:
ex vivo IL6 and IL-10 production of whole blood in response to incubation with E.Coli LPS | 1 day before till 28 days after phlebotomy
  Blood will be drawn on day -1, 0, 1, 3, 5, 7, 14, 21 and 28 after phlebotomy, to assess ex vivo cytokine production.
Changes in hemoglobin, hematocrit, white blood cell count and differential | 1 day before till 28 after phlebotomy
  Hemoglobin, hematocrit, white blood cell count and differential will be determined on day -1, 0, 1, 3, 5, 7, 14, 21 and 28 following the withdrawal of 500 ml of blood at the blood bank
Changes in hemoglobin, hematocrit, white blood cell count and differential | 1 day before till 28 after phlebotomy
  Hemoglobin, hematocrit, white blood cell count and differential will be determined on day -1, 0, 1, 3, 5, 7, 14, 21 and 28 following phlebotomy
Changes in plasma hepcidin | 1 day before till 28 after phlebotomy
  Plasma hepcidin concentration will be determined at various time points during the 28 days of follow-up, following phlebotomy
Changes in other markers of iron homeostasis (serum iron, transferrin saturation, ferritin) | 1 day before till 28 after phlebotomy
  Changes in parameters of iron homeostasis will be determined at various time points during the 28 days of follow-up, following phlebotomy
Adverse Events | 1 day before till 28 after phlebotomy
  Adverse Events will be assessed with every visit

CONTACTS AND LOCATIONS:
Overall Officials: P Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands